CLINICAL TRIAL: NCT04734041
Title: Integrative Medicine for Hypermobility Spectrum Disorder (HSD) and Ehlers-Danlos (EDS) Syndromes: A Mixed-methods Feasibility Study
Brief Title: Integrative Medicine for Hypermobility Spectrum Disorder and Ehlers-Danlos Syndromes (IMforHSDandEDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Healthy Living Community (Unknown)
Responsible Party: Principal Investigator, Douglas Hanes, Associate Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DH10320
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Ehlers-Danlos Syndrome; Hypermobile EDS (hEDS); Hypermobility Syndrome; EDS
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Ehlers-Danlos syndrome type 3 | interventions — Anti-Inflammatory Agents; Diet; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Medicine (Other): Anti-inflammatory (Mediterranean) diet, as well as general behavioral and psychosocial support.
  Interventions: Behavioral: Anti-inflammatory (Mediterranean-style) diet; Behavioral: Behavioral and psychosocial support

INTERVENTIONS:
Behavioral: Anti-inflammatory (Mediterranean-style) diet — Prescription of an anti-inflammatory diet, which encourages increasing whole fruits, vegetables, and grains, as well as balancing macronutrients (proteins, carbohydrates, and fat) for every meal.
Behavioral: Behavioral and psychosocial support — Capture a complete and detailed medical history and background. Discuss familial and social support, provide psychosocial support, assess the patient's current self-management strategies for self-care, and assess the patient's current self-management strategies for mental health. Recommendations will be made in accordance with the needs of the participant.

SUMMARY:
A feasibility study of an integrative medicine program among patients with Hypermobility Spectrum Disorder (HSD) or Ehlers-Danlos syndromes (EDS)

DETAILED DESCRIPTION:
The overall purpose of this study is to assess the feasibility of conducting a 9-week integrative medicine program that is comprised of a prescribed anti-inflammatory (Mediterranean) diet, as well as general behavioral and psychosocial support among patients with Hypermobility Spectrum Disorder (HSD) or Ehlers-Danlos syndromes (EDS), in order to determine the recruitment potential in this population and to measure the ability of individuals to complete the program. Participants will be prescribed a food plan, and adherence to and feasibility of the food plan will be measured through participant food tracking and a subjective assessment of the food plan in a brief satisfaction survey.

This study aims to recruit 20 patients with HSD or EDS and make preliminary observations regarding the effects of integrative medical care on pain reduction and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Beighton score of 4 or more to confirm joint hypermobility diagnosis
* Baseline VAS Score of 1 or more
* Not currently, or already a patient of Dr. Schaefer and Healthy Living Community
* Ability to provide written informed consent
* Willingness to participate in 9-week integrative medicine intervention (and make dietary and lifestyle changes)
* Willingness to attend 1 in-person screening visit and 2 virtual office visits (or 3 virtual visits, if medical documentation of Beighton score can be provided in advance of enrollment, and all other criteria are met)
* Access to an electronic device for MyFitnessPal food-tracker use (i.e mobile device, tablet, laptop)

Exclusion Criteria:

* Pregnant and lactating women, or planned pregnancy over the next 3 months
* Consumption of more than 14 (men) or 7 (women) alcoholic drinks per week
* History of disordered eating or eating disorder
* Body mass index (BMI) considered underweight (<18.5)
* Weight loss from metastatic cancer
* Unable to make dietary changes or participate in a 9-integrative medicine nutritional intervention
* Those with significant dietary changes, new medications, or new exercise routines within the past 90 days
* Currently, or already, a patient of Dr. Schaefer and Healthy Living Community

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 9 weeks
  Number of participants enrolled per month, over the 4 month open recruitment
Retention rate | 9 weeks
  Proportion of participants completing the mid-study or end-of-study visits

SECONDARY OUTCOMES:
Adherence to the dietary recommendations | 5, 9 weeks
  Estimated daily dietary intake recorded in a food tracker app
Adherence to food tracking | 5, 9 weeks
  Reporting per week of dietary intake recorded in a food tracker app

OTHER OUTCOMES:
Visual Analog Scale for Pain (VAS) | Baseline, 5 weeks, 9 weeks
  Baseline, 5-week, and 9-week pain scale scores on a 10-point scale. The numeric measurement of pain between 0 "no pain" and 10 representing "worst pain" will be used.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Baseline, 5 weeks, 9 weeks
  Baseline, 5-week, and 9-week PROMIS pain intensity on a scale of 0 to 10. Higher scores represent greater intensity of pain.
Patient Assessment of Chronic Illness Care (PACIC+) | Baseline, 5 weeks, 9 weeks
  Baseline, 5-week, and 9-week assessment. The PACIC+ consists of 26 items with Likert scale responses on a 5 point scale from "Almost never" to "Almost always," with higher scores representing greater satisfaction with care. The PACIC provides summary scores for attitudes regarding patient-centered care, living with chronic illness, and chronic illness care. All subscales are averages of selected items that range between 1 (poor quality of care received) and 5 (excellent quality of care received).

CONTACTS AND LOCATIONS:
Overall Officials: Rich Barrett, ND, Study Chair — NUNM Institutional Review Board Chair
Locations (2):
- United States (2):
  - National University of Natural Medicine, Portland, Oregon
  - Healthy Living Community, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guedry SE, Langley BO, Schaefer K, Hanes DA. Integrative medicine for hypermobility spectrum disorders (HSD) and Ehlers-Danlos syndromes (EDS): a feasibility study. Disabil Rehabil. 2024 Dec;46(24):5854-5867. doi: 10.1080/09638288.2024.2314713. Epub 2024 Feb 14. PMID 38353245

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04734041/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04734041/ICF_000.pdf